CLINICAL TRIAL: NCT02561468
Title: The Preemptive Analgesic Efficacy of Nefopam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Nefo_breast cancer
Record Dates: First submitted 2015-08-03; First posted 2015-09-28 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — Nefopam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Nefopam (Experimental): 20 mg nefopam in 100 ml normal saline is infused before starting operation.
  Interventions: Drug: Nefopam
- Control (Placebo Comparator): 100 ml normal saline is infused before starting operation.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Nefopam
  Arms: Nefopam
Drug: Saline
  Arms: Control

SUMMARY:
Nefopam is administered as a preemptive analgesic drug to the patient undergoing breast cancer surgery. It will be evaluated whether postoperative acute and chronic pain can be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer
* Lumpectomy with axillary lymph node dissection or Lumpectomy with sentinel lymph node biopsy
* American Society of Anesthesiologists physical status I or II

Exclusion Criteria:

* Refusal
* Seizure
* Cardiac disease
* Monoamine oxidase inhibitor user
* Urologic disease
* Glucoma
* Preoperative analgesic drug medication
* Pregnancy
* Recurred breast cancer patient

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The change of pain numerical rating score from postoperative 30 min until postoperative 3 month | Postoperative 30 min, postoperative 1 day, postoperative 1 week, postoperative 3 month

SECONDARY OUTCOMES:
The dose of ketorolac administered to the patient. | postoperative 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea